CLINICAL TRIAL: NCT01127607
Title: Does Pharmacological Treatment of Attention Deficit Hyperactivity Disorder (ADHD) in Adults Enhance Parenting Performance?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IITWW#2
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: ADHD
Keywords: parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulant medication (Experimental): blinded lisdexamfetamine at the optimal dose for the individual participant as previously determined during the med optimization portion of the study
  Interventions: Drug: lisdexamfetamine
- placebo pill (Placebo Comparator): placebo medication identical in appearance to active med
  Interventions: Drug: lisdexamfetamine

INTERVENTIONS:
Drug: lisdexamfetamine — 3 week with-in subject lead in phase to find optimal dose ranging from 30 mg to 70mg
  Other Names: vyvanse

SUMMARY:
It is now well recognized that Attention-Deficit/Hyperactivity Disorder (ADHD) is a chronic disorder of childhood that extends into adulthood for many individuals. A number of impairments in daily life functioning have been identified in adults with ADHD, including marital distress, risky driving, and using less effective parenting practices (e.g., Barkley, 2006).

Specifically, some parents with ADHD have been found to use inconsistent discipline, less parental involvement, and less positive reinforcement with their children compared to parents without ADHD (e.g., Chen & Johnston, 2007; Chronis-Tuscano, Clarke, Rooney, Diaz, & Pian, 2008). While there is some evidence that stimulant medication improves parental functioning for adults with ADHD, only one study has specifically explored the use of stimulant medication and parenting(Chronis-Tuscano, Seymour, Stine, Jones, Jiles, Rooney, et al., 2008).

The purpose of this study is to explore whether or not the stimulant medication, lisdexamfetamine, improves parent functioning. Measures of parenting behavior, parental psychosocial functioning, and child psychosocial functioning will be collected. It is hypothesized that lisdexamfetamine will be associated with some improvement in these assessments.

DETAILED DESCRIPTION:
Seventy families with at least one parent (either mother or father who will serve as the identified subject) and a school-aged child (ages 5-16) with ADHD will be recruited to participate in a randomized, placebo-controlled trial of lisdexamfetamine to assess the acute and prolonged effects of medication usage on parent-child interactions. The protocol will employ traditional self-report measures of parental competency and functioning used in other studies, but will supplement them with one of the most widely used observational laboratory tasks.

Families will be recruited on a rolling basis and the length of the study will be approximately 8 weeks. In the first three weeks of the study, parents will complete the dose optimization phase to find the optimal dose of lisdexamfetamine. Lisdexamfetamine will be initiated at a dose of 30mg and increased to 50mg for week 2 and 70mg for week 3. During week 4, measures of the acute effects of lisdexamfetamine will be collected, and parents will complete the observational laboratory parent child interaction tasks two times (i.e., on lisdexamfetamine and on placebo- phase I). In the remaining four weeks of the study (phase 2) a between subjects comparison will be conducted. Half of the parents will be randomized to receive lisdexamfetamine and half will receive a placebo. Measures of parent functioning will once again be collected at the end of phase 2 and parents will complete the observational laboratory task, which will allow for exploration of prolonged lisdexamfetamine treatment on parent-child interactions.

ELIGIBILITY:
Inclusion Criteria:

* Parents with a diagnosis of ADHD, who also have a child with an ADHD between the ages of 5-16

Exclusion Criteria:

* Parents with any of the following: any identified structural heart abnormality or other health condition that significantly affects heart performance (e.g., hypertension), a resting systolic blood pressure ≥140 and diastolic blood pressure ≥90, pregnant or breast feeding, significant psychiatric problems other than ADHD that currently require medication or any emergent psychiatric treatment, medical/psychiatric illness that could be worsened by stimulants (such as a seizure disorder, Tourette's Disorder or hyperthyroidism), or alcohol or substance abuse problems in the past 6 months.
* Children with any of the following: any psychiatric problem other than ADHD, Oppositional Defiant Disorder (ODD), or Conduct Disorder (CD) that requires medication or any emergent psychiatric treatment, either parent or child has participated in the same parent-child interaction task used in this study in the last 6 months, either as part of a study or a clinical treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G Waxmonsky, M.D., Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

REFERENCES:
- [Derived] Babinski DE, Waxmonsky JG, Waschbusch DA, Humphery H, Pelham WE Jr. Parent-Reported Improvements in Family Functioning in a Randomized Controlled Trial of Lisdexamfetamine for Treatment of Parental Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2017 Apr;27(3):250-257. doi: 10.1089/cap.2016.0129. Epub 2016 Dec 19. PMID 27991835
- [Derived] Waxmonsky JG, Waschbusch DA, Babinski DE, Humphrey HH, Alfonso A, Crum KI, Bernstein M, Slavec J, Augustus JN, Pelham WE. Does pharmacological treatment of ADHD in adults enhance parenting performance? Results of a double-blind randomized trial. CNS Drugs. 2014 Jul;28(7):665-77. doi: 10.1007/s40263-014-0165-3. PMID 24796970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by direct advertisement as well as from referrals from mental health and medical providers.
Pre-assignment Details: Participants first stabilized on LDX in 3 week open label trial starting at 30mg + increasing by 20mg/week until optimal dose was found. Those unable to tolerate LDX or not responsive to it were discontinued. 38 enrolled; 8 dropped out due to adverse events + 3 were lost to follow up in med phase, leaving 27.
Groups:
- Placebo Arm: All 27 Participants were first optimized on lisdexamfetamine (LDX) (30mg, 50mg or 70mg) over 3 weeks then underwent within-subjects comparison with each subject completed one parent child interaction task (DPICS) once on optimal LDX dose and one parent child interaction task once on placebo (Period 1). The 14 subjects assigned to this arm were then switched to blinded placebo for the parallel group, between subjects trial (period II) which lasted until the final endpoint assessment. These subjects received only placebo during period II.
- Treatment Arm: All 27 Participants were first optimized on lisdexamfetamine (LDX) (30mg, 50mg or 70mg) over 3 weeks then underwent within-subjects comparison with each subject completed one parent child interaction task (DPICS) once on optimal LDX dose and one parent child interaction task once on placebo (Period I). The 13 subjects assigned to this arm were then switched to blinded optimal dose of LDX for the parallel group, between subjects trial (period II) which lasted until the final endpoint assessment. These subjects received only their optimal dose of LDX during period II.
Period: Phase I (Within Subjects)
Arm/Group | Placebo Arm | Treatment Arm
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Phase II (Between Subjects)
Arm/Group | Placebo Arm | Treatment Arm
Started | 14 | 13
Completed | 13 | 11
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adult participant was first stabilized on LDX during a 3 week open label titration. 11 participants dropped out during med titration phase (8 due to adverse events and 3 lost to follow-up; a 12th dropped out after group assignment but prior to receiving blinded phase II medication.
Groups:
- Placebo Arm: Participants in this arm were first optimized on lisdexamfetamine (30mg, 50mg or 70mg) over 3 weeks then switched to blinded placebo for the 4 weeks of the parallel group trial
- Treatment Arm: Participants in this arm were first optimized on lisdexamfetamine (30mg, 50mg or 70mg) over 3 weeks then switched to blinded matching doses of lisdexamfetamine for 4 weeks of the parallel group trial.
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Treatment Arm | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.38 (4.41) | 40.69 (6.06) | 41.04 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Secondary Outcome: Alabama Parenting Questionnaire (APQ)
Description: measures change in parenting practices.The APQ is a 42-item measure (each item ranges from 1/always to 5/never) on which parents are asked to indicate the frequency with which they implement the following parenting practices: involvement (10 items range 10-50- higher scores mean more parental involvement), positive parenting (6 items with range of 6 to 30 and higher scores indicate greater use of praise), poor monitoring/supervision (10 items with range of 10 to 50 and higher scores indicate less supervision/monitoring), inconsistent discipline(6 items with range of 6 to 30 and higher scores indicate greater problems with inconsistent discipline), and corporal punishment (3 items with range of 3-15 and greater scores indicate more use of corporal punishment). Items are rated on a 5-point scale, ranging from 1 ("never") to 5 ("always"). Items summed into composite scales.
  Within subject comparison of no medication baseline vs. optimal dose medication.
Time Frame: baseline and week 4
Population: Used a within-subjects evaluation; the same 24 participants evaluated in both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unmedicated: Data collected at intake, when participants were not on medication
- Optimal Dose of Medication: Data collected after participants received 1 to 3 weeks of their optimal dose of LDX (either 30mg, 50mg or 70mg)
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 24 | 24
units on a scale
  Parent Involvement | 37.83 (5.64) | 38.82 (5.30)
  Positive parenting | 25.42 (3.60) | 25.58 (2.86)
  Poor monitoring and poor supervision | 14.25 (3.84) | 13.58 (3.20)
  Inconsistent discipline | 15.79 (3.51) | 14.62 (3.87)
  Corporal punishment | 4.79 (2.04) | 4.42 (1.72)

2. Secondary Outcome: Disruptive Behavior Disorders Rating Scale (DBD)
Description: Parent ratings of their child's symptoms of attention-deficit hyperactivity disorder (ADHD), oppositional defiant disorder (ODD), and conduct disorder (CD). Measure consists of 45 items each rated on a Likert scale that ranges from 0 (not at all) to 3 (very much). Items are averaged to form adhd-inattention, adhd-hyperactive/impulsive, ODD, and CD scores.Within subject comparison of no medication baseline vs. optimal dose medication. ADHD subscale consists of 20 items with range of 0 to 60. ODD subscale consists of 9 items with range of 0 to 27. CD subscale consists of 15 items with range of 0 to 45. For all subscales, higher scores indicate more severe symptoms.
Time Frame: baseline and week 4
Population: Used a within-subjects design; the same 24 participants measured in both arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 24 | 24
units on a scale
  ADHD-hyperactive/impulsive symptom score | 1.55 (0.76) | 1.34 (0.61)
  ADHD-inattentive symptom score | 2.11 (0.59) | 1.85 (0.74)
  ODD symptom score | 1.17 (0.69) | 1.12 (0.69)
  CD symptom score | 0.16 (0.14) | 0.18 (0.24)

3. Secondary Outcome: Impairment Rating Scale (IRS)
Description: Parent ratings of their child's functioning and need for treatment in developmentally important domains. Ratings are completed using visual-analogue scales that are anchored at the low end by "no problems / no need for treatment" and at the high end by "extreme problem / definitely needs treatment." Visual analogue ratings for each subscale were converted to 0 to 6 scales with higher values indicating greater impairment and lower values indicating less impairment for each subscale.Within subject comparison of no medication baseline vs. optimal dose medication.
Time Frame: baseline and week 4
Population: Uses a within-subjects evaluation; the same 25 participants are in both arms.
Measure: Mean (Standard Deviation); unit: units on a 0 to 6 scale
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 24 | 24
units on a 0 to 6 scale
  Child's peer relationship impairment | 2.75 (2.15) | 2.21 (1.69)
  Child's sibling relationship impairment | 2.82 (2.34) | 2.68 (1.99)
  Child's parent relationship impairment | 3.67 (1.88) | 3.79 (1.56)
  Child's academic impairment | 3.75 (2.13) | 3.29 (2.03)
  Child's self-esteem impairment | 3.92 (1.95) | 3.54 (1.72)
  Child's family impairment | 4.00 (1.83) | 3.87 (1.49)
  Child's overall impairment | 3.63 (1.86) | 3.42 (1.59)

4. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The SDS consists of 3 self rated items assessing the degree to which symptoms affect work/school, social life, and family/home responsibilities. Items are rated on a 0 (not at all) to 10 (extremely) scale. Items were averaged into an overall disability score with range of 0 to 10 with higher scores indicating more severe disability.Within subject comparison of no medication baseline vs. optimal dose medication.
Time Frame: baseline and week 4
Population: Uses a within-subjects design; the same 25 participants are in both arms.
Measure: Mean (Standard Deviation); unit: units on a 0 to 10 scale
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 25 | 25
units on a 0 to 10 scale | 6.26 (2.11) | 3.17 (2.65)

5. Secondary Outcome: Dyadic Parent-Child Interaction Coding System (DPICS)
Description: Observations of parents and children as they interact with each other during a five minute homework task and during a 10 minute non-academic task. Interactions were recorded and later coded by trained observers. Observers counted number of parent and child behaviors with each parent-child dyad counted as one participant. Average number of behaviors per group were computed.This outcome was part of period I- the within subject comparison of all participating subjects once on placebo (n=26) and once with all subjects on active medication (N=26). (the 27th participant completed this phase but partial data was lost due to mechanical failure with video equipment so their data was not included). All adult participants received both placebo and active medication in this phase that comprised all of period 1.
Time Frame: weeks 4 and weeks 5 (period I within subjects trial)
Population: Used a within-subjects design for this phase; the same 26 participants completed all four arms.
Measure: Mean (Standard Deviation); unit: behaviors
Groups:
- Placebo - Homework Task: Parent-child interaction during a homework task. Parents were on placebo and children were unmedicated. Parents and children did not have knowledge of parent treatment condition (medication versus placebo)
- Placebo - Non-academic Task: Parent-child interaction during a non-academic task. Parents were on placebo and children were unmedicated. Parents and children did not have knowledge of parent treatment condition (medication versus placebo)
- Medication - Homework Task: Parent-child interaction during a homework task. Parents were on their optimal dose of lisdexamfetamine (30, 50, or 70 mg) and children were unmedicated. Parents and children did not have knowledge of parent treatment condition (medication versus placebo)
- Medication Non-academic Task: Parent-child interaction during a non-academic task. Parents were on their optimal dose of lisdexamfetamine (30, 50, or 70 mg) and children were unmedicated. Parents and children did not have knowledge of parent treatment condition (medication versus placebo)
Arm/Group | Placebo - Homework Task | Placebo - Non-academic Task | Medication - Homework Task | Medication Non-academic Task
Number analyzed (Participants) | 26 | 26 | 26 | 26
behaviors
  Verbalizations | 61.7 (30.9) | 58.2 (31.1) | 45.2 (21.1) | 48.6 (26.5)
  Commands | 15.4 (11.5) | 14.8 (10.3) | 8.7 (5.2) | 8.3 (4.1)
  inappropriate child behavior | 6.1 (10.0) | 3.3 (4.9) | 2.5 (2.1) | 3.8 (5.4)

6. Secondary Outcome: Dyadic Parent-Child Interaction Coding System (DPICS) - Behavior Percentages
Description: Observations of parents and children as they interact with each other during a five minute homework task and during a 10 minute non-academic task. Interactions were recorded and later coded by trained observers. Observers counted number of parent and child behaviors with each parent-child dyad counted as one participant. Percentages of behaviors as a function of total verbalizations (for praise, negative talk, demanding) or as a function of commands and questions (for impatient and responsive) were computed. This outcome was part of period I- the within subject comparison of all participating subjects once on placebo (n=26) and once with all subjects on active medication (N=26). (the 27th participant completed this phase but partial data was lost due to mechanical failure with video equipment so their data was not included). All adult participants received both placebo and active medication in this phase that comprised all of period 1.
Time Frame: weeks 4 and weeks 5 (period I within subjects trial)
Population: Used a within-subjects design; the same 26 participants completed all arms.
Measure: Mean (Standard Deviation); unit: Percentage of behaviors
Arm/Group | Placebo - Homework Task | Placebo - Non-academic Task | Medication - Homework Task | Medication Non-academic Task
Number analyzed (Participants) | 26 | 26 | 26 | 26
Percentage of behaviors
  Parent praise | 2.6 (3.7) | 3.0 (4.5) | 3.6 (5.8) | 2.2 (2.5)
  Parent negative talk | 4.7 (5.7) | 4.0 (3.6) | 14.4 (11.7) | 9.1 (8.7)
  Parent demandingness | 24.1 (10.7) | 25.7 (11.3) | 19.3 (6.4) | 19.2 (10.5)
  Parent impatient | 39.2 (12.8) | 42.5 (18.7) | 31.2 (15.7) | 32.6 (10.4)
  Parent responsive | 83.2 (25.9) | 74.8 (30.4) | 75.9 (15.3) | 79.8 (12.8)

7. Secondary Outcome: Pittsburgh Side Effect Rating Scale
Description: rates 13 potential adverse events of central nervous system stimulant medications on a 0-3 likert scale with 0=none 1=mild severity, 2=moderate severity, 3=severe severity. Form completed by participants at end of med optimization phase. Mean severity rating then averaged across 13 categories. This compares mean side effect severity at unmedicated baseline state vs. on optimal dose at week 3. Analysis includes all participants completing medication optimization.
Time Frame: baseline and end of dose optimization phase/week 4
Population: Within-subjects analysis; same 26 participants are in the unmedicated and optimal dose of medication arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unmedicated: baseline; participants not on medication
- Optimal Dose of Medication: Optimal dose of lisdexamfetamine (30 mg, 50 mg, or 70 mg) as selected by a three week open medication titration trial.
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 26 | 26
units on a scale | 0.04 (0.12) | 0.26 (0.21)

8. Secondary Outcome: Adult ADHD Rating Scale (ADHD RS)
Description: measures change in all DSM (Diagnostic and Statistics Manual) IV ADHD symptoms on a 0 (least severe) to 3 (most severe) scale. Inattention and hyperactive/impulsive subscales each consist of 9 items with range of 0 to 27. Total Score consists of all 18 items rated 0 to 3 with range of 0 to 54. For all, higher scores indicate more symptoms. All information obtained during clinician interview of patient. At endpoint, the medication group (N=11) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Arm: participants in this arm treated with matching placebo for 4 weeks duration
- Treatment Arm: participants in this arm treated with blinded optimal dose of LDX for 4 weeks (either 30mg, 50mg or 70mg)
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 11
units on a scale
  Inattention | 17.85 (8.21) | 8.82 (6.54)
  Hyperactive/Impulsive | 14.77 (8.23) | 5.64 (5.07)
  Total Score | 32.62 (15.61) | 14.46 (10.91)

9. Secondary Outcome: Parenting Stress Index (PSI)--Total Stress
Description: measures change in stress of parent child interactions and completed by the participant. The PSI is a measure of the source and degree of parenting stress (Abidin, 1995), which contains 120 items which are rated on a 1 (strongly disagree) to 5 (strongly agree) scale. 101 of these items are used to compute a total stress score (reported below) as the other 19 report on specific life stressors. Range is 101 to 505, for which higher scores indicate higher levels of stress. At endpoint, the medication group (N=9) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 9
units on a scale | 241.54 (47.33) | 262.67 (38.84)

10. Secondary Outcome: Parenting Locus of Control (PLC)
Description: self completed parenting measure of the degree to which parents feel they can influence their child's behavior. Measure consists of 25 items each rated using a Likert scales that ranges from 1 ("strongly disagree") to 5 ("strongly agree"). Range is 25 to 125 with higher scores indicating greater parental control over their child's behavior (desired outcome). At endpoint, the medication group (N=9) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 9
units on a scale | 79.00 (4.22) | 80.00 (5.57)

11. Secondary Outcome: Brown Attention Deficit Scale (BAADS)
Description: Measures executive functioning using 40 items each rated using a Likert Scale that ranges from 0 ("never") to 3 ("almost daily"). Activation, Attention and effort subscales are 9 items each with range of 0-27. Affect scale is 7 items (range 0-21), memory is 6 items (range 0-18) and total score is 40 items (range 0-120). All raw scores are then reported as T scores based on normative data with higher T scores indicating worse executive functioning. At endpoint, the medication group (N=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 10
t score
  Activation Scale t-score | 73.38 (11.52) | 66.4 (13.5)
  Attention Scale t-score | 75.54 (11.90) | 65.10 (11.19)
  Effort scale t-score | 72.46 (15.56) | 61.20 (10.98)
  Affect scale t-score | 63.46 (15.37) | 53.20 (5.57)
  Memory scale t-score | 74.38 (63.90) | 13.79 (13.58)
  Total scale t-score | 76.08 (14.79) | 63.30 (70.52)

12. Secondary Outcome: Social Skills Rating System (SSRS)
Description: Measures child's interactions with peers and adults. Items rated using Likert scales that range from 0 ("never") to 2 ("often").At week 8, the medication group (N=10) was compared to the placebo group (N=11). There are two subscales: Problem Behaviors (18 items rated between 0-2 for total score range of 0 to 36) and Social Skills (40 items rated 0-2 with range for total score of 0-80). The total scores for these scales are reported as standard scores, with a population mean of 100 and standard deviation of 15. For problem behavior higher scores indicate worse behavior whereas for social skills, higher scores indicate more social (or better behavior).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: standard scores
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 11 | 10
standard scores
  Social Skills Total Standard Score | 86.64 (17.72) | 89.90 (13.68)
  Problem Behavior Total Standard Score | 113.81 (12.54) | 111.80 (16.55)

13. Secondary Outcome: Disruptive Behavior Disorder Rating Scale (DBD)
Description: measures externalizing symptoms in children.measures externalizing symptoms in children completed by their primary caretaker who was a participant in the study. The DBD (Pelham et al., 1992) assessed DSM symptoms of ADHD, ODD, and CD from 0 (not at all) to 3 (very much). The DBD includes symptoms of DSM-III and DSM-IV ADHD, Oppositional Defiant Disorder (ODD) and Conduct Disorder (CD).At endpoint, the medication group (N=10) was compared to the placebo group (N=12).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 12 | 10
units on a scale
  Inattention | 1.64 (0.76) | 1.60 (0.39)
  Hyperactive/Impulsive | 1.25 (0.66) | 1.09 (0.62)
  Oppositional-defiant | 1.04 (0.56) | 0.76 (0.54)
  Conduct disorder | 0.17 (0.23) | 0.15 (0.16)

14. Secondary Outcome: Impairment Rating Scale (IRS)
Description: measures global functioning of child rated by the parent who was the participant in the study. The IRS is a 7 item measure that uses visual-analogue scales to evaluate the child's problem level and need for treatment in developmentally important areas, such as peer relationships, adult-child relationships, academic performance. Each subscale including overall severity is scored from 0 (no problem) to 6 (extreme problem) with higher scores indicating more impairment. At endpoint, the medication group (N=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 10
units on a scale
  Impairment with peers | 2.62 (2.02) | 2.20 (2.04)
  Impairment with siblings | 2.17 (2.21) | 2.30 (1.89)
  Impairment interferes with parents' relationship | 3.15 (1.57) | 3.10 (1.85)
  Academic impairment | 3.15 (2.23) | 2.60 (2.07)
  Self-esteem impairment | 3.00 (2.04) | 3.40 (1.96)
  General family impairment | 3.08 (1.85) | 2.90 (1.85)
  Overall severity | 2.62 (1.66) | 2.70 (1.64)

15. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The SDS consists of 3 self rated items assessing the degree to which symptoms affect work/school, social life, and family/home responsibilities. Items are rated on a 0 (not at all) to 10 (extremely) scale. Items were averaged into an overall disability score with range of 0 to 10 with higher scores indicating more severe disability. At endpoint, the medication group (N=9) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 9
units on a scale | 4.36 (2.60) | 2.26 (1.90)

16. Secondary Outcome: ADHD Severity Clinical Global Impressions Severity Subscale
Description: clinician rated measure of ADHD symptom severity in adult participants. The severity subscale is scored from 1 (normal) to 7 (extremely ill).At endpoint, the medication group (N=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 11
units on a scale | 3.78 (1.24) | 2.36 (0.81)

17. Secondary Outcome: Barkley Home Situations Questionnaire (HSQ)
Description: Self completed by adult participants. Measures their child's functioning in the evening by asking them to report whether or not their child had problems in developmentally important areas. Number of problems per child are counted and counts are then averaged for each group with higher numbers representing more problems. At endpoint, the medication group (N=9) was compared to the placebo group (N=10).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: number of child problems endorsed
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 10 | 9
number of child problems endorsed | 9.30 (4.67) | 8.67 (5.22)

18. Secondary Outcome: Pittsburgh Side Effect Rating Scale Mean Severity Rating.
Description: rates 13 potential adverse events of Central Nervous System (CNS) stimulants on a 0-3 likert scale with 0=none 1=mild severity, 2=moderate severity, 3=severe severity. Form completed by participants. Mean severity rating then averaged across 13 categories.At endpoint, the medication group (N=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 10
units on a scale | 0.28 (0.10) | 0.26 (0.12)

19. Secondary Outcome: Resting Blood Pressure
Description: Measured at rest at last assessment visit using an automated blood pressure machine; results reported in mmHG. At endpoint, the medication group (N=9) was compared to the placebo group (N=10).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 10 | 9
mm Hg
  systolic BP | 123.40 (8.90) | 122.33 (11.45)
  diastolic BP | 76.10 (8.74) | 75.11 (7.98)

20. Secondary Outcome: Alabama Parenting Questionnaire (APQ)
Description: measures change in parenting practices.The APQ is a 42-item measure (each item ranges from 1/always to 5/never) on which parents are asked to indicate the frequency with which they implement the following parenting practices: involvement (10 items range 10-50- higher scores mean more parental involvement), positive parenting (6 items with range of 6 to 30 and higher scores indicate greater use of praise), poor monitoring/supervision (10 items with range of 10 to 50 and higher scores indicate less supervision/monitoring), inconsistent discipline(6 items with range of 6 to 30 and higher scores indicate greater problems with inconsistent discipline), and corporal punishment (3 items with range of 3-15 and greater scores indicate more use of corporal punishment). Items are rated on a 5-point scale, ranging from 1 ("never") to 5 ("always"). Items summed into composite scales.
  At endpoint, the medication group (N=9) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 9
units on a scale
  Positive parenting | 24.85 (3.46) | 24.33 (3.77)
  Parental involvement | 39.38 (5.38) | 37.78 (4.55)
  Poor monitoring/supervision | 12.23 (3.14) | 12.33 (2.40)
  Inconsistent discipline | 12.46 (3.84) | 14.22 (2.86)
  Corporal punishment use | 4.69 (1.80) | 3.89 (1.17)

21. Secondary Outcome: Impairment Rating Scale (IRS)
Description: self rated measure of global impairment of adult participants derived from the child IRS. The IRS-A assesses impairment overall and in specific domains, including interpersonal relationships, academic performance, and self-esteem, and includes adult-specific domains of functioning, such as employment and romantic relationships. The IRS-A assesses current problems and need for treatment. Each subscale is rated from 0 (no problem) to 6 (extreme problem).At endpoint, the medication group (N=11) was compared to the placebo group (N=13). Overall Impairment is its own subscale and not a composite score of the others.
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 13 | 11
units on a scale
  Impairment with peers | 2.38 (1.50) | 1.91 (1.70)
  Impairment with parents | 2.46 (2.03) | 1.30 (1.64)
  General family impairment | 2.77 (1.88) | 2.27 (1.79)
  Academic impairment | 3.60 (2.88) | 1.83 (2.04)
  Self-esteem impairment | 2.77 (2.09) | 2.00 (1.84)
  Overall impairment | 3.00 (1.73) | 2.55 (1.75)

22. Secondary Outcome: Weight
Description: Weight measured on calibrated scale; participant measured without shoes or heavy clothing (jackets, sweaters, etc...). reported in kilograms.At endpoint, the medication group (N=9) was compared to the placebo group (N=11).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 11 | 9
kg | 76.0 (24.78) | 69.62 (17.71)

23. Primary Outcome: Dyadic Parent-Child Interaction Coding System (DPICS) - Behavior Counts
Description: Observations of parents and children as they interact with each other during a five minute homework task and during a 10 minute non-academic task. Interactions were recorded and later coded by trained observers. Observers counted number of parent and child behaviors. Average number of behaviors per group were computed. Three subjects dropped prior to completing this assessment and one participant completed the other endpoint measures but not the DPICS, which is why the total N for this outcome is 23 at study endpoint. At end of period II (study endpoint), the medication group (n=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Population: Task situation (homework vs. non-academic) was within-subjects; all participants completed both types of interactions. Medication was between subjects.
Measure: Mean (Standard Deviation); unit: behaviors
Arm/Group | Placebo - Homework Task | Placebo - Non-academic Task | Medication - Homework Task | Medication Non-academic Task
Number analyzed (Participants) | 13 | 13 | 10 | 10
behaviors
  Verbalizations | 67.2 (35.4) | 42.1 (16.2) | 53.8 (31.6) | 40.1 (24.0)
  Commands | 14.5 (8.8) | 9.0 (4.2) | 11.0 (6.6) | 4.9 (3.3)
  inappropriate child behavior | 6.8 (6.2) | 1.4 (2.5) | 3.8 (4.7) | 1.5 (1.9)

24. Primary Outcome: Dyadic Parent-Child Interaction Coding System (DPICS) - Behavior Percentages
Description: Observations of parents and children as they interact with each other during a five minute homework task and during a 10 minute non-academic task. Interactions were recorded and later coded by trained observers. Observers counted number of parent and child behaviors. Percentages of behaviors as a function of total verbalizations (for praise, negative talk, demanding) or as a function of commands and questions (for impatient and responsive) were computed.Three subjects dropped prior to completing this assessment and one participant completed the other endpoint measures but not the DPICS, which is why the total N for this outcome is 23 at study endpoint. At end of period II (study endpoint), the medication group (n=10) was compared to the placebo group (N=13).
Time Frame: study endpoint- end of period II (between subjects trial)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Percentage of behaviors
Arm/Group | Placebo - Homework Task | Placebo - Non-academic Task | Medication - Homework Task | Medication Non-academic Task
Number analyzed (Participants) | 13 | 13 | 10 | 10
Percentage of behaviors
  Parent praise | 1.2 (2.2) | 6.0 (6.0) | 2.8 (2.5) | 5.7 (6.2)
  Parent negative talk | 5.3 (4.3) | 5.9 (8.6) | 21.1 (21.0) | 12.6 (10.2)
  Parent demandingness | 21.8 (8.9) | 23.5 (10.9) | 21.7 (10.1) | 12.7 (6.5)
  Parent impatient | 42.4 (11.3) | 38.7 (20.7) | 34.1 (12.9) | 26.3 (11.0)
  Parent responsive | 69.8 (33.3) | 89.7 (18.1) | 63.8 (35.8) | 77.3 (18.8)

25. Secondary Outcome: Resting Pulse
Description: measured at last assessment visit when at rest using an automated blood pressure machine; results reported in beats per minute. At endpoint, the medication group (N=8) was compared to the placebo group (N=9).
Time Frame: study endpoint- end of period II (between subjects trial)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo Arm | Treatment Arm
Number analyzed (Participants) | 9 | 8
bpm | 74.44 (7.58) | 77.13 (4.19)

26. Secondary Outcome: Pittsburgh Side Effects Rating Scale - Percent Present for All Reported Adverse Events Occurring at a Rate of 5% or More
Description: Self report of side effects measured during dose titration using the Pittsburgh Side Effects Rating Scale. Consists of 13 items each rated using 0(none) to 3 (severe) scales. Items endorsed as 1 (mild) or above were counted as present. Information on additional adverse events not part of the PSERS was collected by direct interview of the participants. All side effects occurring at a frequency of 5% or more are reported. Initial side effect data is reported for all participants entering pre-randomization med optimization phase who took medication (n=36) vs those formally enrolled (N=27). Also, side effect data for the med titration phase is entered per dose rather than per participant. For example, a person trying the 30, 50 and 70mg dose is entered is entered 4 times (no med as well) vs. just once. This is why baseline N is higher than for other outcomes collected at weeks 4 and 8 where data was only available for those completing the pre-randomization med optimization phase (N=27).
Time Frame: end of medication optimization phase/week 4
Population: Within-subjects analysis; data entered per dose not per subject. For example, if subject 1 took 30mg, 50mg and 70mgdoses during titration, they are recorded as three separate entries. Sample size reduces as dose increases because participants stopped at lowest acceptable dose and only moved to higher dose if they did not meet optimization criteria.
Measure: Number; unit: Percent of participants
Groups:
- No Medication: The PSERS was completed at intake by all 38 participants who consented and met eligibility criteria in order to assess pre-medication rates of side effects. This was done because the PSERS measures commonly occurring events such as insomnia and irritability that can be seen in unmedicated patients with ADHD.
- 30 mg Lisdexamfetamine: This arm includes all participants who were prescribed the 30mg dose and completed at least one side effect rating for this dose.Not all participants who were prescribed this dose were optimized to this dose or went on to enter the randomized phase of the study which is why this cell size is larger than for the randomized controlled comparison that followed it.
- 50 mg Lisdexamfetamine: This group includes all participants who were prescribed the 50mg dose and completed at least one side effect rating for this dose. All participants reaching this dose were also treated with the 30mg dose and are therefore included in that group as well.Not all participants who were prescribed this dose were optimized to this dose or went on to enter the randomized phase of the study.
- 70 mg Lisdexamfetamine: This group includes all participants who were prescribed the 70mg dose and completed at least one side effect rating for this dose. All participants reaching this dose were also treated with the 30mg and 50mg doses and are therefore included in those groups as well. Not all participants who were prescribed this dose were optimized to this dose.
Arm/Group | No Medication | 30 mg Lisdexamfetamine | 50 mg Lisdexamfetamine | 70 mg Lisdexamfetamine
Number analyzed (Participants) | 38 | 36 | 21 | 17
Percent of participants
  Motor tics | 0 | 0 | 0 | 11.8
  Buccal-lingual movement | 2.6 | 19.4 | 28.6 | 23.5
  picking at skin | 13.2 | 11.1 | 14.3 | 5.9
  worried/anxious | 13.2 | 36.1 | 14.3 | 17.6
  dull, tired, listless | 10.5 | 16.7 | 9.5 | 11.8
  headaches | 5.3 | 36.1 | 28.6 | 29.4
  stomachaches | 0.0 | 16.7 | 4.8 | 29.4
  crabby, irritiable | 10.5 | 27.8 | 23.8 | 23.5
  tearful, sad, depressed | 7.9 | 13.9 | 19.0 | 11.8
  socially withdrawn | 5.3 | 8.3 | 0.0 | 0.0
  loss of appetite | 0.0 | 52.8 | 66.7 | 70.6
  trouble sleeping | 10.5 | 30.6 | 33.3 | 35.3
  dry mouth | 0.0 | 30.6 | 38.1 | 70.5

27. Secondary Outcome: Adult ADHD Rating Scale Completed at the End of the Med Optimization Phase
Description: Measures change in all DSM IV ADHD symptoms on a 0 (least severe) to 3 (most severe) scale. All information obtained during clinician interview of patient. Inattention and hyperactive/impulsive subscales each consist of 9 items with range of 0 to 27. Total Score consists of all 18 items (sum of two subscales) rated 0 to 3 with range of 0 to 54. For all, higher scores indicate more symptoms.
Time Frame: baseline and end of med optimization phase/week 4
Population: Uses a within-subjects design; the same 27 participants are in both arms.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unmedicated | Optimal Dose of Medication
Number analyzed (Participants) | 27 | 27
scores on a scale
  Inattention Symptoms | 23.12 (3.58) | 9.77 (4.44)
  Hyperactive/Impulsive Symptoms | 17.81 (5.73) | 8.00 (5.08)
  Total symptoms | 40.85 (7.55) | 17.77 (8.51)

ADVERSE EVENTS:
Time Frame: Adverse event data reported for period II (mean duration 8 weeks). While 27 total subjects were randomized to a treatment arm (med vs.placebo), 1 withdrew before med was dispensed which is why we have side effect data for 26 and not 27.
Description: Pittsburgh Side Effect Scale (PSERS) was given at every visit to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe). The Columbia-Suicide Severity Rating Scale (C-SSRS) measured suicide risk. It was given at every visit. Both measures were self completed.
Groups:
- Placebo Arm: subjects in this arm treated only with blinded placebo for duration of assessment (period II- between subjects trial).One participant assigned to placebo dropped out before medication was dispensed for period II which is why the side effect data only has a total of 13 and not 14 subjects.
- Treatment Arm: subjects in this arm (N=13) only treated with blinded optimal dose of LDX (either 30mg, 50mg or 70mg) for duration of assessment (period II between subjects trial).
- All Participants in Period 1 Prescribed 30mg: During the dose optimization period which occurred before assignment to the placebo arm or treatment arm, all participants were treated with open label medication starting at 30mg of lisdexamfetamine (LDX). Dose was increased weekly (to a max of 70mg) until the optimal dose was defined. Once optimal dose criteria was met, the titration was stopped. Most participants received multiple doses so results for each dose are presented rather than for each participant.
  All 36 participants who were dispensed the 30mg dose and completed at least one Pittsburgh Side Effect Rating Scale (PSERS) are included in this category.
- All Participants in Period 1 Prescribed 50mg: During the dose optimization period which occurred before assignment to the placebo arm or treatment arm, all participants were treated with open label medication starting at 30mg of lisdexamfetamine (LDX). Dose was increased weekly (to a max of 70mg) until the optimal dose was defined. Once optimal dose criteria was met, the titration was stopped. Most participants received multiple doses so results for each dose are presented rather than for each participant.
  21 of 36 participants were dispensed the 50mg dose.
- All Participants in Period 1 Prescribed 70mg: During the dose optimization period which occurred before assignment to the placebo arm or treatment arm, all participants were treated with open label medication starting at 30mg of lisdexamfetamine (LDX). Dose was increased weekly (to a max of 70mg) until the optimal dose was defined. Once optimal dose criteria was met, the titration was stopped. Most participants received multiple doses so results for each dose are presented rather than for each participant.
  17 of 36 participants were dispensed the 70mg dose.
Arm/Group | Placebo Arm | Treatment Arm | All Participants in Period 1 Prescribed 30mg | All Participants in Period 1 Prescribed 50mg | All Participants in Period 1 Prescribed 70mg
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/36 | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 5/13 | 5/13 | 34/36 | 18/21 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Arm (N=13) | Treatment Arm (N=13) | All Participants in Period 1 Prescribed 30mg (N=36) | All Participants in Period 1 Prescribed 50mg (N=21) | All Participants in Period 1 Prescribed 70mg (N=17)
suicidal ideation (Psychiatric disorders) | 0 (0) | 0/11 (0) | 0 (0) | 0 (0) | 0 (0) — Every participant completed the Columbia Suicide Severity Rating Scale (CSSRS) at each visit. It assess suicidal ideation and self harm attempts including preparatory and interrupted attempts.
self harm attempt (Psychiatric disorders) | 0 (0) | 0/11 (0) | 0 (0) | 0 (0) | 0 (0) — Measured at each visit using the self completed CSSRS.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=13) | Treatment Arm (N=13) | All Participants in Period 1 Prescribed 30mg (N=36) | All Participants in Period 1 Prescribed 50mg (N=21) | All Participants in Period 1 Prescribed 70mg (N=17)
Buccal Lingual Movements (Nervous system disorders) | 2 (2) | 0 (0) | 7 (7) | 6 (6) | 4 (4) — Pittsburgh Side Effect Scale (PSERS):Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
picking at skin (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 1 (1) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
anxious/jittery (Psychiatric disorders) | 3 (3) | 3 (3) | 13 (13) | 3 (3) | 3 (3) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
fatigue (General disorders) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 2 (2) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
headache (Nervous system disorders) | 0 (0) | 1 (1) | 13 (13) | 6 (6) | 5 (5) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
irritability (Psychiatric disorders) | 1 (1) | 3 (3) | 10 (10) | 5 (5) | 4 (4) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 2 (2) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
appetite decrease (General disorders) | 2 (2) | 3 (3) | 19 (19) | 14 (14) | 12 (12) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
insomnia (General disorders) | 4 (4) | 3 (3) | 11 (11) | 7 (7) | 6 (6) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This event was spontaneously reported. It is not listed on the PSERS.
dry mouth (Endocrine disorders) | 1 (1) | 3 (3) | 11 (11) | 8 (8) | 12 (12) — This event was spontaneously reported. It is not listed on the PSERS.refers to participants report of experiencing decreased salivation or a sense of "dry mouth"
stomachache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 5 (5) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
socially withdrawn (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).
motor tic (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Pittsburgh Side Effect Scale (PSERS) was given at baseline and endpoint to all participants to measure adverse events. It contains 13 items measured medication side effects from 0 (none) to 3 (severe).

LIMITATIONS AND CAVEATS:
This study was limited by its small sample size. The validity and psychometrics of DPICS in adolescents is not well established, but removal of the adolescents had little impact on study results and actually strengthened some observed effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No